CLINICAL TRIAL: NCT00004353
Title: Study of the Metabolism of Pyruvate and Related Problems in Patients With Lactic Acidemia
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of California, San Diego (Other)
Other Study IDs: NCRR-M01RR00827-0071; UCSD-071
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2008-07-10 (Estimated); Status verified 2002-04

CONDITIONS: Mitochondrial Myopathy; MELAS Syndrome; Lactic Acidosis
Keywords: MELAS syndrome; inborn errors of metabolism; lactic acidosis; mitochondrial myopathy; rare disease
MeSH Terms: conditions — Mitochondrial Myopathies; MELAS Syndrome; Acidosis, Lactic; Metabolism, Inborn Errors; Rare Diseases

SUMMARY:
OBJECTIVES: I. Study the metabolism of pyruvate and related problems in patients with lactic acidemia.

II. Define the nature of the metabolic defect.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients fast for 6 hours. Glucagon IM is administered after the 6 hour fast. Glucose level is measured at 0, 15, 30, 45, 60, and 90 minutes.

In children of sufficient size, alanine and lactic acid should also be measured at each or most of these time points.

Fasting continues for at least 18 hours. Glucagon IM is administered again at end of fast. Glucose level is measured at time 0, 15, 30, 45, 60, and 90 minutes.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

* Diagnostically documented elevation in lactate, pyruvate, and/or alanine levels in lactic acidemia patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 1978-12

CONTACTS AND LOCATIONS:
Overall Officials: Richard H. Haas, Study Chair — University of California, San Diego
Locations (1):
- University of California San Diego Medical Center, San Diego, California, United States